CLINICAL TRIAL: NCT02225197
Title: A Phase II Study of Fractionated CyberKnife Stereotactic Radiosurgery to Perioptic Tumors
Brief Title: A Phase II Trial of CyberKnife Radiosurgery to Perioptic Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Cancer Center, Normal, Illinois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK Perioptic-01
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Tumor, Benign, Optic Nerve
Keywords: Perioptic; Stereotactic; Radiation; Benign brain tumor; Optic apparatus
MeSH Terms: conditions — Optic Nerve Neoplasms; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CyberKnife Radiosurgery (Experimental)
  Interventions: Radiation: CyberKnife Radiosurgery

INTERVENTIONS:
Radiation: CyberKnife Radiosurgery — 25 Gy delivered in 5 fractions of 5 Gy per fraction
  Other Names: CyberKnife

SUMMARY:
The purpose of this study is to find out what effects (good and bad) CyberKnife stereotactic radiosurgery has on tumors near the critical structures of the eye (optic apparatus).

The investigators hypothesize that hypofractionated stereotactic radiotherapy via the CyberKnife ® can deliver tumor ablating doses of radiation to perioptic lesions safely and effectively while sparing the adjacent optic apparatus and normal brain tissues from receiving damaging doses of radiation.

DETAILED DESCRIPTION:
The CyberKnife system is a type of radiation machine that uses a special system to precisely focus large doses of x-rays (radiation) on the tumor. The device is designed to concentrate large doses of radiation onto the tumor so that injury from radiation to the nearby normal tissue will be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Perioptic lesion within 2mm of the optic apparatus
* Age >= 21
* KPS >= 50
* Planning Target Volume (PTV) <= 6.0 cm in maximal diameter

Exclusion Criteria:

* Malignant histology
* Age < 21
* KPS <= 40
* Planning Target Volume (PTV) > 6.0 cm in maximal diameter
* Prior whole brain XRT
* Gross total resection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Tumor status | 5 years
  To determine the local control rate of patients with perioptic lesions treated with stereotactic CyberKnife radiosurgery.

CONTACTS AND LOCATIONS:
Overall Officials: Shermian Woodhouse, MD, Principal Investigator — Community Cancer Center
Locations (1):
- Community Cancer Center, Normal, Illinois, United States